CLINICAL TRIAL: NCT03948282
Title: Ultrasound Assessment of the Inferior Vena Cava in Children; Comparison of Sub-xiphoid and Right Lateral Coronal Views During Spontaneous Ventilation
Brief Title: Ultrasound Assessment of the Inferior Vena Cava in Children
Status: Completed | Type: Observational
Sponsor: Alok Moharir (Other)
Responsible Party: Sponsor-Investigator, Alok Moharir, Pediatric Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00000316
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, non-blinded observational study to compare measurement of inferior vena cava (IVC) dimensions with two placement sites of the ultrasound probe (sub-xiphoid and the side or right lateral position).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 patients scheduled for elective dental surgery under general anesthesia.

Exclusion Criteria:

* History of significant pulmonary disease, cardiac disease, and laparotomy.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing elective dental surgery.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
IVC diameter | Baseline
  Measurement of the inferior vena cava via ultrasound using the right lateral view and the subxiphoid view.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States